CLINICAL TRIAL: NCT03352739
Title: A Randomized Controlled Study of 12 Months to Evaluate the Safety and Efficacy of Deep Brain Stimulation(DBS) to the Fornix & Meynert Nucleus(NbM) in Patients With Mild to Moderate Alzheimer's Disease(AD)
Brief Title: Fornix and NbM as Targets of Stimulation In Alzheimer's Disease
Acronym: FANTASIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XuanwuH
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- DBS of the fornix, power on (Experimental)
  Interventions: Device: DBS of the fornix, power on
- DBS of the NbM, power on (Experimental)
  Interventions: Device: DBS of the NbM, power on
- DBS of the fornix, power off (Sham Comparator)
  Interventions: Device: DBS of the fornix, power off
- DBS of the NbM, power off (Sham Comparator)
  Interventions: Device: DBS of the NbM, power off
- Control group (No Intervention): The patients are going to prescribe stable dosage of donepezil during observation period without surgical interference.

INTERVENTIONS:
Device: DBS of the fornix, power on — DBS of bilateral columns of the fornix is performed, with the power of the device on since the 1st month after the implantation. Observations will start at the time when the device is turning on .
  DBS system includes:
  Pins G102 Implantable Neurostimulator; Pins L301 DBS Electrode； Pins E202 DBS extension lead
  Arms: DBS of the fornix, power on
Device: DBS of the NbM, power on — DBS of bilateral NbMs is performed, with the power of the device on since the 1st month after the implantation. Observations will start at the time when the device is turning on .
  DBS system includes:
  Pins G102 Implantable Neurostimulator; Pins L301 DBS Electrode； Pins E202 DBS extension lead
  Arms: DBS of the NbM, power on
Device: DBS of the fornix, power off — DBS of bilateral columns of the fornix is performed, the power of the device is going to keep off during the first 7 months after the implantation. Observations will start after 1 month of the implantation.
  DBS system includes:
  Pins G102 Implantable Neurostimulator; Pins L301 DBS Electrode； Pins E202 DBS extension lead
  Arms: DBS of the fornix, power off
Device: DBS of the NbM, power off — DBS of bilateral NbMs is performed, the power of the device is going to keep off during the first 7 months after the implantation. Observations will start after 1 month of the implantation.
  DBS system includes:
  Pins G102 Implantable Neurostimulator; Pins L301 DBS Electrode； Pins E202 DBS extension lead
  Arms: DBS of the NbM, power off

SUMMARY:
The primary goal of this study is to evaluate the efficacy and safety of the DBS to the fornix/NbM among patients who are diagnosed as AD according to a series of evaluations including cerebrospinal fluid (CSF) biomarkers and molecular imaging examinations; The secondary goal is to compare the efficacy among the two treatment groups of different targets.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with informed consent;
2. 45-75 years of age;
3. At least 6 years of education;
4. AD according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) guidelines (McKhann et al., 2011);
5. Clinical Dementia Rating Scale (CDR): 1.0-2.0;
6. Positive findings with amyloid PET imaging;
7. Stable prescription of donepezil (5mg, qd) for at least 3 months, and without any intentions to modify the dosage during the observation period.

Exclusion Criteria:

1. Fazekas scale>2;
2. Neuropsychiatric inventory (NPI) total score ≥10, or any subdomain≥4；
3. Modified Hachinski ischemic score>4；
4. Young Mania Rating Scale>11(Young, Biggs, Ziegler, & Meyer, 1978);
5. Any suicidal tendencies in recent 2 years;
6. Cornell Scale for Depression and Dementia>10;
7. Familial AD;
8. Abnormal brain structural magnetic resonance imaging (MRI) scan, including hydrocephalus, stroke, structural lesions, etc. that would potentially confound the outcome;
9. Surgical history of the central nervous system;
10. Severe cardiovascular/pulmonary disorders.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive outcome | 12 months (from 1 month to 13 month after implantation)
  Cognitive function measured by Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-cog, 13-items version).
  ADAS-cog 13 scale range: 0-80; (Higher value represents a worse outcome)

SECONDARY OUTCOMES:
Neuroplasticity outcome | 12 months (from 1 month to 13 month after implantation)
  Protection of hippocampal volume revealed by magnetic resonance imaging (MRI).
Neuroplasticity outcome | 12 months (from 1 month to 13 month after implantation)
  Improved cerebral metabolic level revealed by FDG positron emission tomography(PET) imaging.
Cognitive outcome | 12 months (from 1 month to 13 month after implantation)
  Improvement of cognitive function evaluated by Clinical Dementia Rating Scale sum of the boxes (CDR-SB).
  CDR-SB scale range: 0-18; ("0" represents normal cognition, the higher the score, the worse the cognitive function).
Functional outcome | 12 months (from 1 month to 13 month after implantation)
  Improvement of life quality according to Activities of Daily Living (ADL) scale.
  ADL scale range: 20-80 ("20" represents normal life ability, the higher the score, the worse the life ability).
Safety outcome | 12 months (from 1 month to 13 month after implantation)
  Device/therapy related side effects or complications such as mortality an morbidity.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China